CLINICAL TRIAL: NCT02318485
Title: Translational Stem Cell Research in Ophthalmology - Regenerating the Anterior Cornea Through Standardized Transplantation of Limbal Epithelial Stem Cells: a Phase II Multicenter Trial
Brief Title: Limbal Epithelial Stem Cell Transplantation: a Phase II Multicenter Trial
Acronym: MLEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRG13-003
Record Dates: First submitted 2014-12-02; First posted 2014-12-17 (Estimated); Last update posted 2025-01-15 (Actual); Status verified 2024-06

CONDITIONS: Limbal Stem Cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

ARMS (1):
- Transplant (Experimental): A limbal epithelial stem cell graft will be transplanted onto the limbal stem cell deficient eye after it has been debrided of fibrovascular pannus
  Interventions: Biological: Limbal epithelial stem cell graft

INTERVENTIONS:
Biological: Limbal epithelial stem cell graft
  Other Names: limbo-amnion composite graft; Limbal stem cell graft

SUMMARY:
This project aims to conduct a multicentre human clinical trial to effectively diagnose and treat limbal stem cell deficiency (LSCD) which can be caused by a number of different disease processes, all of which have a common denominator, i.e. a loss of the normal functioning epithelial stem cells of the cornea. A number of different diseases such as aniridia, steven johnson's syndrome, ocular cicatricial pemphigoid, bacterial keratitis, or chemical and thermal injuries to the cornea can lead to gradual loss of its functioning epithelial stem cells. This leads to vascularization of the cornea with surrounding conjunctival epithelium growing over it resulting in its scarring and opacification. These corneas, since vascular, no longer retain their immune privilege and prove extremely challenging to the ophthalmic surgeon. Grafting donor corneas which in normal circumstances (non vascular corneas) would give excellent results, exhibit high rates of rejection. This can be very frustrating for both the patient as well as the surgeon. Since there are a number of different contributing disease pathologies, our estimate is that there are approximately 100 patients per year in Belgium that suffer from some degree of LSCD. These patients are very often not correctly diagnosed since this is a relatively new disease first described in 1990 after the discovery of limbal epithelial stem cells in 1989. The low rates of diagnosis could potentially be increased by in vivo confocal scanning microscopy as a non invasive screening test to detect early signs of LSCD and therefore offer conservative treatment options. In the cases where total limbal stem cell deficiency has already developed, conventional corneal grafting is not suitable due to the high vascularity of the host bed. In this situation we propose transplanting standardized limbal epithelial stem cell grafts generated from the patient's own ocular stem cells (from the good eye, where available) or from HLA matched donors. Tiny 1 by 2mm superficial limbal (peripheral cornea) biopsy can be taken and the epithelial stem cells expanded in the laboratory on a biological substrate, until there is a graft measuring >8mm in diameter generated in 2 a week period. This can then be transplanted onto the diseased eye after removal of scar tissue using a novel surgical technique we have developed.

DETAILED DESCRIPTION:
This project aims to conduct a multicenter, single-arm phase II study, in which we will assess the safety and efficacy of transplanting standardized, non-xenogenic limbal stem cell grafts for patients with LSCD. The Good Manufacturing Practice (GMP) clean room facilities at the Centre for Cell Therapy and Regenerative Medicine (CCRG, UZA) will conduct tissue engineering, while the Departments of Ophthalmology at the University Hospitals in Antwerp (UZA), Brussels (UZB) and Gent (UZG) will enrol patients, perform pre-operative tests, harvest the limbal biopsies, perform the auto- or allogenic graft transplantation and follow-up. Based on the past experience from our phase I/II mono-centre human clinical trial, we have been able to document the safety and feasibility of the transplantation. 12/18 patients (2/3 allogenic and 10/15 autologous) have shown decrease in corneal vascularization, complete epithelialization and incorporation of the graft into the anterior cornea post limbal stem cell transplantation. However our current results are limited with respect to the sample size, feasibility of allogenic transplantation (only 3 cases), long term follow-up (mean of 22 months, range 4-43 months) and disease monitoring strategies. Longer patient follow-up to determine long term success (especially following subsequent corneal transplants) and inclusion of a larger allogenic patient population need to be addressed before this treatment can be translated to the clinics and recognized by the RIZIV as a reimbursable cell therapy.

It is pertinent to say that this cell based therapy has the potential to provide this orphan pathology with an effective treatment option. The Flemish society will benefit from this project by improved rehabilitation of patients suffering from corneal blindness due to LSCD. By providing this treatment option we can offer a ray of hope to patients that would formerly have to learn to live with their disability. By restoring vision for these patients it is possible to reintegrate them into society as socially accepted individuals. Even a small degree of visual rehabilitation can make all the difference. For example, a slight increase in visual acuity can restore a person's ability to drive rather than having them rely exclusively on public transportation. More independence and a better quality of life are the main objectives that we are striving to achieve as the major outcome of this project.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years
2. Voluntary written informed consent
3. Patients suffering from LSCD IIa and IIb. Those suffering from IIc may be included once inflammation has subsided and cornea can be staged as IIb.
4. Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
5. Women of child-bearing potential should use adequate contraception prior to study entry and for the duration of study participation. Negative serum or urine β-HCG pregnancy test at screening.

Exclusion Criteria:

1. Subjects who are pregnant or lactating
2. Subjects who have sensitivity to drugs that provide local anesthesia
3. Subjects suffering from active infection of the external eye
4. Medical conditions that prohibit the use of systemic immunosuppression (in cases of allogenic transplantation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2023-01 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
Visual acuity | one year
  using Log MAR scale
presence of persistent epithelial defects | 3 months post surgery
  using Fluorescein drops and cobalt blue filter photography at the slit lamp
presence of corneal conjunctivalization | one year
  slit lamp photography and in vivo confocal microscopy
change in corneal vascularization | one year
  slit lamp photography
Eye pain | one year
  using visual pain scale
photophobia | one year
  using a 4 point scale
Rejection | one year
  Increased neovascularization, epithelial defects and a drop in visual acuity Redness Pain Irritation slit lamp examination

CONTACTS AND LOCATIONS:
Overall Officials: Sorcha Ni Dhubhghaill, Principal Investigator — University Hospital, Antwerp
Locations (3):
- Belgium (3):
  - Antwerp University Hospital, Edegem, Antwerp
  - University Hospital Brussels, Brussels
  - University Hospital, Ghent, Ghent

REFERENCES:
- [Result] Zakaria N, Possemiers T, Dhubhghaill SN, Leysen I, Rozema J, Koppen C, Timmermans JP, Berneman Z, Tassignon MJ. Results of a phase I/II clinical trial: standardized, non-xenogenic, cultivated limbal stem cell transplantation. J Transl Med. 2014 Mar 3;12:58. doi: 10.1186/1479-5876-12-58. PMID 24589151